CLINICAL TRIAL: NCT01385111
Title: Combined Application of EBUS-TBNA and EUS-B-FNA in Mediastinal Staging of Lung Cancer; EBUS-TBNA Centered Procedure vs. EUS-B-FNA Centered Procedure, a Randomized Study.
Brief Title: Combined Application of EBUS and EUS in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Bin, Hwangbo, National Cancer center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NCC-EUSEBUS
Record Dates: First submitted 2011-06-23; First posted 2011-06-29 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2011-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: endobronchial ultrasound; endoscopic ultrasound; EBUS-TBNA; EUS-FNA; EUS-B-FNA; lung cancer; staging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): EBUS centered
  Interventions: Procedure: EUS-B-FNA followed by EBUS-TBNA
- Arm B (Experimental): EUS centered
  Interventions: Procedure: EBUS-TBNA followed by EUS-B-FNA

INTERVENTIONS:
Procedure: EUS-B-FNA followed by EBUS-TBNA — EUS-B-FNA will be performed followed by EBUS-TBNA when additional needle aspiration is necessary after EBUS-TBNA.
  Arms: Arm A
Procedure: EBUS-TBNA followed by EUS-B-FNA — EBUS-TBNA will be performed followed by EUS-B-FNA when additional needle aspiration is necessary after EUS-B-FNA
  Arms: Arm B

SUMMARY:
This study aims to investigate a diagnostic yield and performance characteristics according to the order of endobronchial ultrasound guided transbronchial needle aspiration (EBUS-TBNA) and endoscopic ultrasound-with bronchoscope-guided transbronchial needle aspiration (EUS-B-FNA) in the mediastinal staging of potentially operable lung cancer. EUS-FNA is a better tolerated procedure than EBUS-TBNA. Therefore, EUS-B-FNA can be the main procedure in a combined approach with EBUS-TBNA and EUS-B-FNA. In group A, the investigators perform EBUS-TBNA first and EUS-B-FNA is performed when necessary. In group B, EUS-B-FNA is first applied and EBUS-TBNA is performed when necessary. The hypothesis is that the diagnostic yield of the EUS centered procedure is as good as that of the EBUS centered procedure and the EUS centered procedure is more tolerable than the EBUS centered procedure. We evaluate diagnostic yields and performance characteristics of each group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or strongly suspected non-small cell lung cancer (NSCLC)
* Potentially operable patients

Exclusion Criteria:

* M1 disease
* Inoperable T4 disease
* Mediastinal infiltration or extranodal invasion of the mediastinal lymph node visible on chest CT.
* Confirmed supraclavicular lymph node metastasis
* Pancoast tumors
* Medically inoperable patients
* Contraindications for bronchoscopy and esophageal endoscopy
* Drug reaction to lidocaine, midazolam,fentanyl
* Pregnancy
* Ground glass-dominant nodule ( < 3cm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | When the confimative disgnosis is available in all subjects (after surgery) ; 8-12 months

SECONDARY OUTCOMES:
Procedure time | During and just after the procedure ; 5-60 minutes
Cardiovascular measurement (change of blood pressure, changes of heart rate, number of patients with arrhythmia) | During the procedure; 0-60 minutes
Degree of desaturation | During the procedure; 0-60minutes
Discomfort by the procedure | After the procedure ; 2-3hr
Number of participants with adverse Events (infection, bleeding requiring intervention, pneumothorax, or any complications requiring hospital admission) | During and after the procedure; 0-2 weeks
Lymph node features | During and after the procedure; 0-2hrs
Fentanyl/midazolam/lidocaine consumption | After the procedure ; 1-2 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Bin Hwangbo, MD, PhD, Principal Investigator — Medical Doctor, Senior Researcher
Locations (1):
- National Cancer Center (NCC) Korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kang HJ, Hwangbo B, Lee GK, Nam BH, Lee HS, Kim MS, Lee JM, Zo JI, Lee HS, Han JY. EBUS-centred versus EUS-centred mediastinal staging in lung cancer: a randomised controlled trial. Thorax. 2014 Mar;69(3):261-8. doi: 10.1136/thoraxjnl-2013-203881. Epub 2013 Oct 30. PMID 24172712